CLINICAL TRIAL: NCT05688579
Title: Effect of Mineralcorticoid Recept Antagonist on Cardiovascular Disease in Patients With Hypertension and Hyperaldosteronemia：A Multicenter Randomized Controlled Study
Brief Title: Effect of MRA on Cardiovascular Disease in Patients With Hypertension and Hyperaldosteronemia
Acronym: EMRACHH
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Li (Other)
Responsible Party: Sponsor-Investigator, Nanfang Li, Professor, Chief physician, People's Hospital of Xinjiang Uygur Autonomous Region
Organization: People's Hospital of Xinjiang Uygur Autonomous Region (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A.HT.2022.8.4
Record Dates: First submitted 2023-01-05; First posted 2023-01-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Hypertension; Hyperaldosteronaemia
MeSH Terms: conditions — Hypertension; Hyperaldosteronism | interventions — Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mineralocorticoid Receptor Antagonists(MRAs) (Experimental): Participants will treat with mineralocorticoid receptor antagonists(MRAs) (including spironolactone 20-60mg/ day, or eplerenone50-100mg/day, or finerenone 10-20mg/ day) in addition to the original antihypertensive drugs for 48 months.
  Interventions: Drug: Mineralocorticoid Receptor Antagonists(MRAs)
- Blank Control (Placebo Comparator): Participants will be given the original antihypertensive drugs for 48 months.
  Interventions: Other: Blank control

INTERVENTIONS:
Drug: Mineralocorticoid Receptor Antagonists(MRAs) — Participants will be treated with mineralocorticoid receptor antagonists(MRAs) in addition to the original antihypertensive drugs for 48 months.
  Arms: Mineralocorticoid Receptor Antagonists(MRAs)
Other: Blank control — Participants will be treated with the original antihypertensive drugs for 48 months.
  Other Names: Placebo
  Arms: Blank Control

SUMMARY:
Elevated aldosterone causes moderate to severe increase in blood pressure, and leads to various target organ damage including cardiovascular ones. Aldosterone has been considered one of the important risk factors for cardiovascular and cerebrovascular diseases. Currently, the use of mineralocorticoid receptor antagonists(MRA) has been proven to reduce blood pressure levels, but long-term prognostic data are lacking in hypertensive patients. Therefore, the purpose of this clinical trial is to assess the effect of MRA on cardiovascular disease in patients with Hypertension and Hyperaldosteronemia.

DETAILED DESCRIPTION:
The trial will randomize about 7800 participants aged between 30 and 75 years with Hypertension and Hyperaldosteronemia(Plasma aldosterone concentration >12 ng/dl). All participants were randomly assigned to two different intervention groups. One group was treated with mineralocorticoid receptor antagonists(MRAs) (including spironolactone 20-60mg/ day, or eplerenone50-100mg/day, or finerenone 10-20mg/ day) in addition to the original antihypertensive drugs. One group was given the original antihypertensive drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old;
2. Blood pressure ≥140/90 mmHg, or have taken antihypertensive drugs;
3. Plasma aldosterone concentration> 12ng/ dL;
4. Serum potassium < 4.8mmol/L;
5. Signed the written informed consent.

Exclusion Criteria:

1. SBP/DBP≥190/120mmHg, DBP<60 mmHg;
2. Known secondary cause of hypertension, including pheochromocytoma, primary aldosteronism (adrenal tumor > 1cm), Cushing's syndrome, renal artery stenosis, renin tumor, connotation of aorta, etc.;
3. History of ischemic or hemorrhagic stroke within the last 3 months (not lacunar infarction and transient ischemic attack [TIA]).
4. History of Hospitalization for myocardial infarction or unstable angina, or coronary revascularization (PCI or CABG) within the last 3 months.
5. History of aortic dissection/dissection aneurysm rupture.
6. History of NYHA Grade III-IV heart failure or hospitalization Aggravated chronic heart failure upon admission within the last 3 months.
7. A history of persistent atrial fibrillation, atrial flutter, or other severe arrhythmias on admission (including sinus delay, diseased sinus, high atrioventricular block, frequent ventricular morning, etc.).
8. Severe liver disease or liver dysfunction: AST, ALT, or ALP > 5ULN (5 times the upper limit of normal), or BIL > 3ULN (3 times the upper limit of normal).
9. End-stage renal disease (ESRD) on dialysis, or estimated glomerular filtration rate (eGFR) <30 mL/min, or serum creatine >2.5 mg/dl [>221 umol/L];
10. Patients with serious physical diseases such as malignant tumors and autoimmune diseases.
11. Severe cognitive or mental impairment.
12. Pregnant and lactating women.
13. Those who have contraindications or allergies to MRAs.
14. Patients with hypoadrenocortical function.
15. Participating in other clinical trials.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of the composite endpoint | 4 years
  A composite endpoint comprised of occurrence of symptomatic stroke ( ischemic or hemorrhagic stroke), acute coronary syndrome (myocardial infarction and hospitalization for unstable angina), hospitalization for decompensated heart failure, coronary revascularization (percutaneous coronary intervention [PCI], coronary artery bypass grafting [CABG]), atrial fibrillation, aortic dissection and dissection aneurysm, and death from cardiovascular causes.

SECONDARY OUTCOMES:
Occurrence of symptomatic stroke ( ischemic or hemorrhagic) | 4 years
  Stroke is defined as a rapid onset of focal (or global) disturbance of cerebral function lasting more than 24 hours (except interrupted by surgery or death) without resolution of symptoms according to the World Health Organization. The diagnosis of stroke is confirmed by strict neurological examination, computed tomography (CT), or magnetic resonance imaging (MRI), and stroke subtypes are classified including ischemic or hemorrhagic, fatal or not fatal.
Occurrence of cardiac adverse events(Acute coronary syndrome and coronary revascularization) | 4 years
  Acute coronary syndrome includes myocardial infarction and hospitalization for unstable angina. The diagnosis of MI is based on the following criteria: (1) Patient has cardiac signs and symptoms, such as retrosternal pain last for at least 30 minutes, and not relieve to nitroglycerine during the attack; (2) Electrocardiographic abnormal findings of MI are observed; (3) Biochemical markers of cardiac damage are present.The diagnosis of unstable angina requires hospitalization for evaluation. The clinical presentation of unstable angina includes: (1) prolonged (>20 min) angina pain at rest; (2) new onset angina; (3) post-MI angina; (4) recent destabilization of previously stable angina with at least Canadian Cardiovascular Society Class III angina characteristics. Patients are treated with coronary revascularization by either PCI or CABG due to acute coronary syndromes (ACS) and stable ischemic heart disease (SIHD).
Occurrence of aortic dissection and dissection aneurysm | 4 years
  Aortic dissection and dissection aneurysms are diagnosed based on basic information, blood biochemical information and imaging information.
Occurrence of Hospitalization for acute decompensated heart failure | 4 years
  Diagnosis of acute decompensated heart failure requires a hospitalization or emergency department visit which provides an infusion therapy for clinical signs and symptoms consistent with cardiac decompensation or inadequate cardiac pump function, such as increasing or new onset shortness of breath, peripheral edema, paroxysmal dyspnea, orthopnea, or hypoxia.
Occurrence of Atrial fibrillation | 4 years
  Diagnosis of AF requires rhythm evidence of an ECG showing the typical pattern including absolutely irregular RR intervals and no discernible, distinct P waves.
Occurrence of all-cause death | 4 years
  All-cause death includes death due to any reasons during the trial. Evidence for death includes death certificates from hospitals or reports of home visit from investigators.
Occurrence of Decline in renal function or development of end stage renal disease (ESRD) | 4 years
  Decline in renal function is assessed by any of the following: (1) For patients with chronic kidney disease (eGFR <60 ml per minute per 1.73 m2) at baseline, the renal outcome was a composite of a decrease in the eGFR of 50% or more (confirmed by a subsequent laboratory test) or the development of ESRD requiring long-term dialysis or kidney transplantation; or (2) For participants without chronic kidney disease at baseline, the renal outcome was defined by a decrease in the eGFR of 30% or more to a value of less than 60 ml per minute per 1.73 m2.
First occurrence of diabetes mellitus | 4 years
  Diagnosis of incident diabetes mellitus includes the following criteria: (1) Fasting plasma glucose ≥ 126 mg/dl (≥ 7.0 mmol/dl); or (2) Oral glucose tolerance test 2-hour glucose in venous plasma ≥ 200 mg/dl (≥ 11.1 mmol/l); or (3) In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥ 200 mg/dl (≥ 11.1 mmol/l); or (4) Glycosylated hemoglobin (HbA1c) ≥ 6.5% (48 mmol/mol).
First occurrence of nonalcoholic fatty liver | 4 years
  Diagnosis of nonalcoholic fatty liver disease includes the following criteria: (1) imaging or histological evidence of hepatic steatosis; (2) Except other causes of secondary fat accumulation in the liver.
Occurrence of Decline in cognitive function | 4 years
  Decline in cognitive function includes sensory disturbance, memory disorders and thinking disorders, which is assessed by mini-mental state examination (MMSE).
Changes in vascular elasticity from baseline（ABI and baPWV） | 1-4 years
  Ankle brachial index [ABI],and brachial-ankle pulse wave velocity(baPWV) well-established non-invasive techniques for evaluating obstruction and stiffness of peripheral artery respectively, are considered for the purposes of cardiovascular risk assessment. ABI is the ratio of the average systolic blood pressure measured in brachial/ankle, and an ABI between and including 0.9 and 1.2 is considered normal, while a lesser than 0.9 indicates arterial disease. The unit measure of baPWV value is cm per second.
Changes in urine protein from baseline | 1-4 years
Changes in cardiac structural indicators from baseline | 1-4 years
  Ventricular septal thickness and left ventricular posterior wall thickness were evaluated mainly by echocardiography.
Blood pressure control rate | 1-3months
  Blood pressure control was assessed by home blood pressure or ambulatory blood pressure for 7 consecutive days

CONTACTS AND LOCATIONS:
Locations (1):
- Hypertension Center of People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaclavik J, Sedlak R, Plachy M, Navratil K, Plasek J, Jarkovsky J, Vaclavik T, Husar R, Kocianova E, Taborsky M. Addition of spironolactone in patients with resistant arterial hypertension (ASPIRANT): a randomized, double-blind, placebo-controlled trial. Hypertension. 2011 Jun;57(6):1069-75. doi: 10.1161/HYPERTENSIONAHA.111.169961. Epub 2011 May 2. PMID 21536989
- [Result] Monticone S, D'Ascenzo F, Moretti C, Williams TA, Veglio F, Gaita F, Mulatero P. Cardiovascular events and target organ damage in primary aldosteronism compared with essential hypertension: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2018 Jan;6(1):41-50. doi: 10.1016/S2213-8587(17)30319-4. Epub 2017 Nov 9. PMID 29129575
- [Result] Williams B, MacDonald TM, Morant S, Webb DJ, Sever P, McInnes G, Ford I, Cruickshank JK, Caulfield MJ, Salsbury J, Mackenzie I, Padmanabhan S, Brown MJ; British Hypertension Society's PATHWAY Studies Group. Spironolactone versus placebo, bisoprolol, and doxazosin to determine the optimal treatment for drug-resistant hypertension (PATHWAY-2): a randomised, double-blind, crossover trial. Lancet. 2015 Nov 21;386(10008):2059-2068. doi: 10.1016/S0140-6736(15)00257-3. Epub 2015 Sep 20. PMID 26414968
- [Result] Cannone V, Buglioni A, Sangaralingham SJ, Scott C, Bailey KR, Rodeheffer R, Redfield MM, Sarzani R, Burnett JC Jr. Aldosterone, Hypertension, and Antihypertensive Therapy: Insights From a General Population. Mayo Clin Proc. 2018 Aug;93(8):980-990. doi: 10.1016/j.mayocp.2018.05.027. PMID 30077215
- [Result] Joseph JJ, Echouffo-Tcheugui JB, Kalyani RR, Yeh HC, Bertoni AG, Effoe VS, Casanova R, Sims M, Wu WC, Wand GS, Correa A, Golden SH. Aldosterone, Renin, Cardiovascular Events, and All-Cause Mortality Among African Americans: The Jackson Heart Study. JACC Heart Fail. 2017 Sep;5(9):642-651. doi: 10.1016/j.jchf.2017.05.012. Epub 2017 Aug 16. PMID 28822744
- [Result] Inoue K, Goldwater D, Allison M, Seeman T, Kestenbaum BR, Watson KE. Serum Aldosterone Concentration, Blood Pressure, and Coronary Artery Calcium: The Multi-Ethnic Study of Atherosclerosis. Hypertension. 2020 Jul;76(1):113-120. doi: 10.1161/HYPERTENSIONAHA.120.15006. Epub 2020 May 18. PMID 32418495
- [Result] Ni X, Zhang J, Zhang P, Wu F, Xia M, Ying G, Chen J. Effects of spironolactone on dialysis patients with refractory hypertension: a randomized controlled study. J Clin Hypertens (Greenwich). 2014 Sep;16(9):658-63. doi: 10.1111/jch.12374. Epub 2014 Jul 22. PMID 25052724